CLINICAL TRIAL: NCT04711057
Title: CENTR(AR): Lungs Moving
Acronym: CENTR(AR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Programa Operacional Inclusão Social e Emprego (POISE) (Unknown); Programa Operacional Competitividade e Internacionalização (POCI) - Compete2020 (Unknown); Portuguese National Funding Agency for Science, Research and Technology (FCT) (Unknown); Aveiro Institute of Biomedicine (iBiMED) (Unknown); School of Health Sciences, University of Aveiro (ESSUA) (Unknown); City Council/Municipality: a) Aveiro; b) Estarreja; c) Oliveira do Bairro; d) Montemor-o-Velho (Unknown); Administração Regional de Saúde do Centro, IP (ARS Centro) (Unknown); Centro Hospitalar do Baixo Vouga (CHBV), E.P.E. (Unknown)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Associate Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POISE-03-4639-FSE-000597
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Chronic Respiratory Disease; Lung Diseases; Pulmonary Disease; Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease
Keywords: Chronic Respiratory Disease; Pulmonary Rehabilitation; Physical Activity; Behavioral Change
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Rehabilitation + Community-based PA program (Experimental): After PR, the experimental group will integrate a community-based PA program.
  Interventions: Other: Community-based PA program; Other: Pulmonary Rehabilitation
- Pulmonary Rehabilitation (Active Comparator): The control group will only receive pulmonary rehabilitation, which integrates PA recommendations.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Community-based PA program — After completing the PR program, the experimental group (EG) will enroll in a 6-month personalized community-based PA program, which should be attended twice-weekly, minimum. During the first month the physiotherapist will guide patients through all available physical activities; afterwards, patients will be asked to choose one or two activities, according to their preference, which they'll attend for five more months. Physiotherapists' support will gradually decrease over time.
  Arms: Pulmonary Rehabilitation + Community-based PA program
Other: Pulmonary Rehabilitation — Exercise training, twice a week, and education and psychosocial support once every other week during 12 weeks.

SUMMARY:
Chronic Respiratory Diseases (CRDs) are associated with substantial morbidity and mortality, ranking as the third leading cause of death worldwide. Pulmonary rehabilitation (PR) is a fundamental evidence-based intervention for the management of a variety of CRDs, such as Chronic Obstructive Pulmonary Disease (COPD) and Interstitial Lung Diseases (ILDs). However, the benefits of PR tend to decline over time and there is currently no strong evidence that patients translate those benefits into a more active lifestyle. There is an urgent need for evidence-based interventions to promote physical activity (PA) participation, whilst maintaining PR positive effects in the long-term. Community-based PA interventions adjusted to the local context, as well as patients' needs and preferences, might be a key strategy to meet this target. CENTR(AR) will be a sustainable response to support healthy lifestyles and enhance long-term PR benefits, by providing access to PR within Primary Healthcare Centres (PHC), followed by the inclusion in a community-based PA program, which embraces urban facilities and available resources.

DETAILED DESCRIPTION:
The Global Burden Disease Study 2017 estimated that 544.9 million people worldwide had a chronic respiratory disease (CRD). Globally, it is estimated that 3.914.196 deaths were due to CRDs in 2017, accounting for 7% of total all-cause deaths, ranking CRDs as the third leading cause of death worldwide. Pulmonary rehabilitation (PR) is a well-established, cost-effective intervention for the management of CRDs (e.g., COPD, ILD), which has been found to improve exercise capacity, dyspnoea and quality of life. Unfortunately, PR remains an underutilized resource in the community. Despite substantial improvement following PR, benefits tend to decline over time (approximately, within a 12-month period) and there is currently no strong evidence that patients translate those benefits into a more active lifestyle. This is of utmost importance since physical activity (PA) levels predict important outcomes in COPD, for example, with low PA levels being associated with a higher risk of exacerbation-related hospitalization and mortality. That said, it is still unknown how best to maintain long-term effects of PR, whilst promoting patients' adherence to a physically active lifestyle. Most studies reporting on interventions to improve PA among patients with CRDs (e.g., COPD) focus exclusively on patients' individual factors, disregarding interpersonal/social and environmental factors associated with PA. Community-based PA interventions adjusted to the local context, which leverage existing social support and community (infra)structures, may be key elements for success. Indeed, the community offers a variety of physical activity modalities (e.g., urban trails, physical activity/exercise classes at the municipality level), which can be explored and further personalized to meet patients' needs and preferences. By targeting the community, as opposed to the "individual per se", the possibility of promoting a behavioral change towards a more physically active lifestyle becomes more likely. Building on existing knowledge, CENTR(AR) primary aim is to implement and assess the effectiveness of a personalised community-based PA program to increase PA levels, as well as prevent/stop the decline and consolidate PR benefits (in several health-related domains) in people with CRDs, following PR.

Additionally, CENTR(AR) will also aim at:

1) Improving access to and delivery of community-based PR for people with CRDs in Primary Healthcare Centres (PHC) within the Centre Region of Portugal; 2) Identifying barriers and facilitators, as well as preferences and motivations of adherence to PA; 3) Educating/Empowering/Capacitating non-health professionals delivering municipal physical activity/exercise classes, to ensure patients' safety and quality care; 4) Designing and validating urban walking and/or cycling trails by a) measuring the physiological response and energy expenditure associated with the use of those trails; b) assessing the environmental/physical features of the urban trails; 5) Validating the available municipal physical activity/exercise classes (as described in 3); 6) Promoting intersectoral collaboration at the municipality level, leveraging partnerships between PHC and existing community physical activities, thereby filling in the gaps in the continuity of care after PR; 7) Increasing health literacy amongst municipal professionals in regard to CRDs, as well as health promotion and community empowerment.

Randomized Controlled Trial (RCT)

Aims & Outcomes Primary aim: Assess the effectiveness of a community-based PA program, tailored to patient's needs and preferences, to increase PA levels in people with CRDs.

Secondary aim(s): Determine the short-, mid- and long-term effects of CENTR(AR) on exercise capacity, functional status, HRQoL, symptoms, AECOPD and healthcare utilisation, peripheral muscle strength, motivation for exercise, and emotional status; Establish the influence of patients' motivations and preferences in adhering to the CENTRAR program and engaging in a physically active lifestyle.

At each time-point, the following data will be collected: Socio-demographic and anthropometric data; Lung function; Healthcare utilization; Health-related quality of life (HRQoL); Impact of disease; Fatigue; Dyspnoea; Cough and sputum; Social support and social network; Anxiety and depression; Motivation to exercise; Perception of change; Exercise capacity; Peripheral muscle strength; Functional status; Balance; Physical activity levels; Adverse events; Adherence; Qualitative data (individual and focus groups interviews)

Study Design & Intervention

After completion of PR, participants will be randomised to an experimental group (EG) or a control group (CG). The EG will enrol in a 6-month personalised community-based PA program, which will/should be attended twice-weekly, minimum. During the first month the physiotherapist will guide patients through all available physical activities; afterwards, patients will be asked to choose one or two activities, according to their preferences, which they will attend for five more months. Physiotherapists' support will gradually decrease over time. The CG will receive a leaflet with PA recommendations.

Sample Size Estimation

The sample size was estimated using G*Power 3.1.9.6, with an effect size specification "as in G*Power 3.0", for the within-between interaction of a repeated measures ANOVA with two groups (control and experimental) and 3 measurements (immediately after, and 6 to 12 months post-PR) of the defined primary outcome (MVPA). The investigators considered an α of 0.05, a power of 0.80, a repeated measures correlation of 0.5, a nonsphericity correction of 1 and an expected effect size f of 0.30. The effect size f was derived from the partial η2 of 0.21 (f=0.516) obtained from a study which aimed to assess the impact of a PA-focused behavioural intervention during and after PR on PA levels in patients with COPD. A smaller f value of 0.30 was chosen to account for a longer follow-up period (up to 12 months) and differences in selected time-points. The calculated sample size was 20 (i.e., 10 in each group) COPD patients and considering a possible 50% dropout rate, the final sample size was determined to be 40. Since no significant differences are expected in the primary outcome between COPD and ILD patients, a sample size of 40 was also determined for the latter. In summary, a total sample size of 80 was found to be required to detect significant within-between group differences in MVPA.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a chronic respiratory disease;
* Stable clinical condition (defined as no acute exacerbation or hospitalization in the previous month).

Exclusion Criteria:

* Signs of cognitive impairment;
* Neoplasic/Immunologic disease or an unstable/significant cardiac (e.g., exertional angina, valvular heart disease, congestive heart failure, etc.), musculoskeletal/orthopaedic, neuromuscular or psychiatric condition limiting ability to exercise or co-operate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in PA levels (time spent in moderate to vigorous physical activity (MVPA)) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Time spent in MVPA will be collected with the ActiGraph accelerometry-based activity monitors (wGT3X-BT) during for week. Raw data will be downloaded, summed and filtered by the ActiLife software (Version 6.13.4) to determine the average MVPA (min/wk).

SECONDARY OUTCOMES:
Change in PA levels (time spent in sedentary behaviour) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Time spent in sedentary behaviour will be collected with the ActiGraph accelerometery-based activity monitors (wGT3X-BT) for one week. Raw data will be downloaded, summed and filtered by the ActiLife software (Version 6.13.4).
Change in step count (steps/day-1) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Steps/day-1 will be collected with the ActiGraph accelerometery-based activity monitors (wGT3X-BT) for one week. Raw data will be downloaded, summed and filtered by the ActiLife software (Version 6.13.4).
Change in health-related quality of life (HRQoL) - St. George Respiratory Questionnaire | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  The St. George Respiratory Questionnaire (SGRQ) will be used to measure disease-specific impact on overall health, daily life and perceived well-being. The SGRQ is standardized self-administered 50-item questionnaire divided into three subscales: symptoms (eight items), activity (sixteen items) and impact (twenty-six items). Scores range from 0 to 100, with higher scores indicating more limitations.
Change in exercise capacity/tolerance - 6-minute walk test (6MWT) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  The 6MWT is a sub-maximal exercise test used to assess (aerobic) exercise capacity that entails measurement of distance walked over a total of 6 minutes (back and forth a 30-m indoor, unobstructed, flat, straight enclosed corridor.) Distance covered will be recorded in metres.
Change in overall functional status/physical function - Physical Performance Test | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Functional status will be assessed with the Physical Performance Test, which comprises multiple domains of physical function using tasks that replicate activities of daily living (ADLs). This measure has 9-items with a total score of 36 points, with higher scores indicating better performance.
Change in quadriceps muscle strength - Isometric dynamometry | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Quadriceps muscle strength will be measured using a hand-held dynamometer (kilogram/force).
Change in handgrip strength - Isometric dynamometry | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Handgrip strength will be measured with a hand-held dynamometer (kilogram)
Healthcare utilisation - AECOPD frequency (previous year) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Number of exacerbations the year prior will be collected, since exacerbation rate/frequency is associated with accelerated lung function decline.
Healthcare utilisation - Emergency department visits (number of visits per participant) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Healthcare utilization will be assessed through the number of emergency department visits per participant the year prior.
Change in healthcare utilization - Hospital (re)admissions (number of hospital admissions per participant) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Healthcare utilization will be assessed through the number of hospital admissions each participant had in the previous year.
Change in healthcare utilization - Hospital (re)admissions (length of stay per hospital admission) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Healthcare utilization will be assessed by the average of days that patients spent in the hospital (length of stay), per admission, in the previous year.
Change in motivation to exercise - The Behavioural Regulation Exercise Scale-2 (BREQ-2) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  The Behavioural Regulation Exercise Scale-2 (BREQ-2) will be used to assess behavioural regulation according to self-determination theory (SDT) relative to exercise participation. A 5-point Likert scale, ranging from 0 = "Not True" to 4 = "Very true", is used to rate each of its 18 items. The items are grouped into six subscales (amotivation, external regulation, introjected regulation, identified regulation, integrated regulation and intrinsic motivation), which reflect the motivational continuum of SDT.
Change in PA levels - Brief Physical Activity Questionnaire | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  The Brief Physical Activity Questionnaire will be used to assess patients' PA. The Brief PA-tool consists of 2 questions assessing the frequency and duration of time spent in moderate to vigorous PA (MVPA) in a 'usual' week. A total score is calculated (0-8). If the sum of the 2-item scores is above or equal to 4 the subject will be considered physically active.
Change in impact of symptoms - COPD Assessment Test (CAT) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  COPD Assessment Test (CAT) consists of 8 items assessing various manifestations/symptoms of COPD (cough, sputum, dyspnoea, chest tightness, confidence, activity, sleep and energy levels) aiming to provide quantified measure of health status. CAT scores range from 0-40; higher scores denote a more severe impact of COPD on patients' lives.
Change in emotional status - Hospital Anxiety and Depression Scale (HADS) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  Hospital Anxiety and Depression Scale (HADS) will be used to assess symptoms of anxiety and depression. It is a 14-item questionnaire that can be subdivided in two subscales: anxiety and depression. Scores are provided for each subscale and range from 0 to 21, with higher scores meaning more symptoms of anxiety and depression.
Change in subjective experience of fatigue - Checklist of Individual Strength - Fatigue subscale | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  The Checklist of Individual Strength (CIS-FS) - Fatigue subscale will be used to assess subjective experience of fatigue. The CIS-FS consists of 8 items with a 7 point-Likert scale scoring. A total score is derived by summation of the item scores.
Change in impact of fatigue - Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  The Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-F) is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function. A 5-point Likert-type scale is used to rate each of the 13 items. The score range is 0 to 52, with 0 being the worst possible score and 52 being the best possible score indicating no fatigue.
Change in impact of cough and sputum - Cough and Sputum Assessment Questionnaire (CASA-Q) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  The CASA-Questionnaire will be used to assess the impact of cough and sputum on patients' lives. The CASA-Q is a 20-item, 5-point rating scale, composed of 4 domains (cough symptoms; cough impact; sputum symptoms; sputum impact) - three (items) per each symptom domain, and eight and six in the cough and sputum impact domains, respectively.
Change in exercise tolerance/capacity and (lower limb) functional capacity - 1-minute sit-to-stand test | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  The patient is seated upright on a chair of standard height of 46 cm, without arm rests, positioned against a wall. The patient sat with the knees and hips flexed to 90°, feet placed flat on the floor hip-width apart, and hands placed on the hips. Subjects are asked to perform repetitions of standing upright and sitting down, as many times as possible at a self-paced speed for one minute, without using their arms for support while rising or sitting.
Change in perceived social support - six-item Social Support Questionnaire (SSQ6) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  A Portuguese-version of the Social Support Questionnaire - Short-Form (SSQ-6), a brief 6-question/item version of the original 27-item questionnaire, will be used to assess the availability and satisfaction of a person's social support.
Change in peripheral muscle strength (one- (1RM) or ten- (10RM) repetition maximum) | before PR (T0), immediately after PR (T1), and after a 3, 6 and 12 month-period.
  The one-repetition maximum (1RM) method, defined as the maximal weight that can be lifted once with correct lifting technique, will be used to a) measure/determine (peripheral) muscle strength and b) derive strength/resistance training intensity. In alternative to 1RM, the result of multiple repetition testing (10RM) will be used to predict/estimate the one-repetition maximum.
Quality trail experience | Immediately after PR
  Participants outdoor experience will be assessed in a small group of patients. They will be asked to participate in an interview whilst taking one of the urban/rural trails adapted to people with chronic lung disease, to collect, for example, user's perception of the trail environment and recreation experience and make adjustments informed by their perceptions.
Adherence to the physical activity programme | Adherence will be collected in each session of physical activity throughout the 6 months.
  Participants from the EG adherence to the physical activity programme will be registered by the sports professional responsible for each physical activity and by participants' using a diary
Occurrence of adverse events | Occurrence of an adverse event will be collected in each session of physical activity throughout the 6 months
  The occurrence of adverse events in the EG during the physical activity programme will be registered by the sports professional responsible for each physical activity and by participants' in their diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S. Marques, PhD, Principal Investigator — School of Health Sciences, University of Aveiro (ESSUA)
Locations (1):
- School of Health Sciences of the University of Aveiro (ESSUA), Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD Chronic Respiratory Disease Collaborators. Prevalence and attributable health burden of chronic respiratory diseases, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Respir Med. 2020 Jun;8(6):585-596. doi: 10.1016/S2213-2600(20)30105-3. PMID 32526187
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944
- [Background] Dowman L, Hill CJ, Holland AE. Pulmonary rehabilitation for interstitial lung disease. Cochrane Database Syst Rev. 2014 Oct 6;(10):CD006322. doi: 10.1002/14651858.CD006322.pub3. PMID 25284270
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Spruit MA, Pitta F, McAuley E, ZuWallack RL, Nici L. Pulmonary Rehabilitation and Physical Activity in Patients with Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2015 Oct 15;192(8):924-33. doi: 10.1164/rccm.201505-0929CI. PMID 26161676
- [Background] Gimeno-Santos E, Frei A, Steurer-Stey C, de Batlle J, Rabinovich RA, Raste Y, Hopkinson NS, Polkey MI, van Remoortel H, Troosters T, Kulich K, Karlsson N, Puhan MA, Garcia-Aymerich J; PROactive consortium. Determinants and outcomes of physical activity in patients with COPD: a systematic review. Thorax. 2014 Aug;69(8):731-9. doi: 10.1136/thoraxjnl-2013-204763. Epub 2014 Feb 20. PMID 24558112
- [Background] Burge AT, Cox NS, Abramson MJ, Holland AE. Interventions for promoting physical activity in people with chronic obstructive pulmonary disease (COPD). Cochrane Database Syst Rev. 2020 Apr 16;4(4):CD012626. doi: 10.1002/14651858.CD012626.pub2. PMID 32297320
- [Background] Mantoani LC, Rubio N, McKinstry B, MacNee W, Rabinovich RA. Interventions to modify physical activity in patients with COPD: a systematic review. Eur Respir J. 2016 Jul;48(1):69-81. doi: 10.1183/13993003.01744-2015. Epub 2016 Apr 21. PMID 27103381
- [Background] Robinson H, Williams V, Curtis F, Bridle C, Jones AW. Facilitators and barriers to physical activity following pulmonary rehabilitation in COPD: a systematic review of qualitative studies. NPJ Prim Care Respir Med. 2018 Jun 4;28(1):19. doi: 10.1038/s41533-018-0085-7. PMID 29867117
- [Background] Arbillaga-Etxarri A, Gimeno-Santos E, Barberan-Garcia A, Balcells E, Benet M, Borrell E, Celorrio N, Delgado A, Jane C, Marin A, Martin-Cantera C, Monteagudo M, Montella N, Munoz L, Ortega P, Rodriguez DA, Rodriguez-Roisin R, Simonet P, Toran-Monserrat P, Torrent-Pallicer J, Vall-Casas P, Vilaro J, Garcia-Aymerich J. Long-term efficacy and effectiveness of a behavioural and community-based exercise intervention (Urban Training) to increase physical activity in patients with COPD: a randomised controlled trial. Eur Respir J. 2018 Oct 18;52(4):1800063. doi: 10.1183/13993003.00063-2018. Print 2018 Oct. PMID 30166322
- [Background] Cruz J, Brooks D, Marques A. Walk2Bactive: A randomised controlled trial of a physical activity-focused behavioural intervention beyond pulmonary rehabilitation in chronic obstructive pulmonary disease. Chron Respir Dis. 2016 Feb;13(1):57-66. doi: 10.1177/1479972315619574. Epub 2015 Dec 23. PMID 26703921
- [Background] Wootton SL, Hill K, Alison JA, Ng LWC, Jenkins S, Eastwood PR, Hillman DR, Jenkins C, Spencer LM, Cecins N, McKeough ZJ. Effects of Ongoing Feedback During a 12-Month Maintenance Walking Program on Daily Physical Activity in People with COPD. Lung. 2019 Jun;197(3):315-319. doi: 10.1007/s00408-019-00216-5. Epub 2019 Apr 15. PMID 30982940
- [Background] Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7. doi: 10.1016/s0954-6111(06)80166-6. PMID 1759018
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Reuben DB, Siu AL. An objective measure of physical function of elderly outpatients. The Physical Performance Test. J Am Geriatr Soc. 1990 Oct;38(10):1105-12. doi: 10.1111/j.1532-5415.1990.tb01373.x. PMID 2229864
- [Background] O'Shea SD, Taylor NF, Paratz JD. Measuring muscle strength for people with chronic obstructive pulmonary disease: retest reliability of hand-held dynamometry. Arch Phys Med Rehabil. 2007 Jan;88(1):32-6. doi: 10.1016/j.apmr.2006.10.002. PMID 17207672
- [Background] Markland, D. and V. Tobin, A Modification to the Behavioural Regulation in Exercise Questionnaire to Include an Assessment of Amotivation. 2004. 26(2): p. 191.
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Crawford B, Monz B, Hohlfeld J, Roche N, Rubin B, Magnussen H, Nivens C, Ghafouri M, McDonald J, Tetzlaff K. Development and validation of a cough and sputum assessment questionnaire. Respir Med. 2008 Nov;102(11):1545-55. doi: 10.1016/j.rmed.2008.06.009. Epub 2008 Jul 27. PMID 18662868
- [Background] Ozalevli S, Ozden A, Itil O, Akkoclu A. Comparison of the Sit-to-Stand Test with 6 min walk test in patients with chronic obstructive pulmonary disease. Respir Med. 2007 Feb;101(2):286-93. doi: 10.1016/j.rmed.2006.05.007. Epub 2006 Jun 27. PMID 16806873
- [Background] Sarason, I.G., et al., A Brief Measure of Social Support: Practical and Theoretical Implications. Journal of Social and Personal Relationships, 1987. 4(4): p. 497-510.